CLINICAL TRIAL: NCT01893554
Title: A Phase I Study of the Safety and Immunogenicity of a Single Dose of the Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine RSV ΔNS2 Δ1313 I1314L, Lot RSV#006A, Delivered as Nose Drops to RSV-Seropositive Children 12 to 59 Months of Age, RSV-Seronegative Infants and Children 6 to 24 Months of Age, and Infants 4 to 6 Months of Age
Brief Title: Evaluating the Safety and Immune Response to a Single Dose of a Respiratory Syncytial Virus (RSV) Vaccine in Infants and Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 288; CIR 288 (Other: WIRB)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group 1: RSV vaccine (Experimental): Healthy RSV-seropositive children ages 12 to 59 months will receive one dose of the RSV ΔNS2 Δ1313 I1314L vaccine administered as nose drops at study entry.
  Interventions: Biological: RSV ΔNS2 Δ1313 I1314L Vaccine
- Group 1: Placebo (Placebo Comparator): Healthy RSV-seropositive children ages 12 to 59 months will receive one dose of the placebo administered as nose drops at study entry.
  Interventions: Biological: Placebo
- Group 2: RSV vaccine (Experimental): Healthy RSV-seronegative infants and children ages 6 to 24 months will receive one dose of the RSV ΔNS2 Δ1313 I1314L vaccine administered as nose drops at study entry.
  Interventions: Biological: RSV ΔNS2 Δ1313 I1314L Vaccine
- Group 2: Placebo (Placebo Comparator): Healthy RSV-seronegative infants and children ages 6 to 24 months will receive one dose of the placebo administered as nose drops at study entry.
  Interventions: Biological: Placebo
- Group 3: RSV vaccine (Experimental): Healthy RSV-seronegative infants and children ages 6 to 24 months will receive one dose of the RSV ΔNS2 Δ1313 I1314L vaccine administered as nose drops at study entry.
  Interventions: Biological: RSV ΔNS2 Δ1313 I1314L Vaccine
- Group 3: Placebo (Placebo Comparator): Healthy RSV-seronegative infants and children ages 6 to 24 months will receive one dose of the placebo administered as nose drops at study entry.
  Interventions: Biological: Placebo
- Group 4: RSV vaccine (Experimental): Healthy infants between the ages 4 to 6 months who have not been screened for RSV serostatus will receive one dose of the RSV ΔNS2 Δ1313 I1314L vaccine administered as nose drops at study entry.
  Interventions: Biological: RSV ΔNS2 Δ1313 I1314L Vaccine
- Group 4: Placebo (Placebo Comparator): Healthy infants between the ages 4 to 6 months who have not been screened for RSV serostatus will receive one dose of the placebo administered as nose drops at study entry.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV ΔNS2 Δ1313 I1314L Vaccine — For participants in Groups 1, 3, and 4: 10^6 plaque forming units (PFU) of RSV ΔNS2 Δ1313 I1314L vaccine will be administered as nose drops (0.25 mL per nostril for a total of 0.5 mL).
  For participants in Group 2: 10^5 PFU of RSV ΔNS2 Δ1313 I1314L vaccine will be administered as nose drops (0.25 mL per nostril for a total of 0.5 mL).
  Arms: Group 1: RSV vaccine; Group 2: RSV vaccine; Group 3: RSV vaccine; Group 4: RSV vaccine
Biological: Placebo — Placebo will be administered as nose drops (0.25 mL per nostril for a total of 0.5 mL).
  Arms: Group 1: Placebo; Group 2: Placebo; Group 3: Placebo; Group 4: Placebo

SUMMARY:
Human respiratory syncytial virus (RSV) is a common cause of respiratory illness in infants and children around the world. This study will evaluate the safety and immune response to a RSV vaccine in three groups of participants: healthy children who have already had an RSV infection (RSV seropositive), healthy infants and children who have not already had an RSV infection (RSV seronegative), and healthy younger infants who have not been screened for prior RSV infection.

DETAILED DESCRIPTION:
RSV is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age around the world. RSV illness can range from mild upper respiratory tract illness (URI) to severe LRI, including bronchiolitis and pneumonia. The purpose of this study is to evaluate the safety and immunogenicity of a single dose of a RSV vaccine in healthy children. Study researchers will first evaluate the vaccine in healthy RSV-seropositive children, then evaluate the vaccine in healthy RSV-seronegative infants and children, followed by younger infants not screened for RSV serostatus.

This study will first enroll healthy RSV-seropositive children ages 12 to 59 months (Group 1). At study entry, participants will undergo a medical history review, physical examination, blood collection, and a nasal wash procedure. Participants will be randomly assigned to receive either the RSV vaccine or placebo vaccine, administered as nose drops. Subjects will be actively monitored for 28 days following administration of vaccine or placebo; monitoring will include medical history reviews, clinical assessments, and at some visits, nasal washes. On the days where no study visit is scheduled, study researchers will contact participants' parents or guardians for medical follow-up.

Study researchers will evaluate the study data of participants in Group 1 before enrolling participants in Group 2, and study data from Group 2 will be reviewed before enrolling participants in Group 3. Finally, study data from Group 3 will be reviewed before enrolling participants in Group 4. Participants in Groups 2 and 3 will include healthy RSV-seronegative infants and children ages 6 to 24 months. Participants in Group 4 will include healthy infants, ages 4 to 6 months, who have not been screened for RSV serostatus.

Participants in Groups 2, 3, and 4 will be randomly assigned to receive either the RSV vaccine or placebo vaccine, administered as nose drops. Subjects will be actively monitored for 56 days following administration of vaccine or placebo; monitoring will include medical history reviews, clinical assessments, and at some visits, nasal washes. On the days where no study visit is scheduled, study researchers will contact participants' parents or guardians for medical follow-up. At a study visit on Day 56, participants will undergo a medical history review, blood collection, and a nasal wash procedure.

For participants in Groups 2, 3, and 4, from November through March following each participant's vaccination visit, parents or guardians will monitor participants for RSV-associated illnesses and report these on a weekly basis via telephone calls to study researchers. Participants may have additional study visits that may include blood collection and/or nasal wash procedures during this follow-up period. Participants in Groups 3 and 4 will have the option to take part in additional monitoring for a second RSV season.

ELIGIBILITY:
Inclusion Criteria for Seropositive Children:

* Healthy children at least 12 but less than 60 months of age, whose parent/guardian understands and signs the study informed consent and who agrees to vaccine administration following a detailed explanation of the study
* Seropositive for RSV as defined by serum RSV neutralizing antibody titer equal to or greater than 1:40. If a child at least 12 but less than 60 months of age is determined to be RSV seropositive prior to Day 56, s/he does not need an additional screening serum specimen, but a pre-inoculation serum specimen must be obtained.
* Participant's history has been reviewed and participant has undergone a physical examination indicating that s/he is in good health
* Participant is expected to be available for the duration of the study

Exclusion Criteria for Seropositive Children:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy including systemic corticosteroids, or bone marrow/solid organ transplant recipients (topical steroids, topical antibiotics, and topical antifungal medications are acceptable)
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an RSV vaccine or previous receipt of or planned administration of any anti-RSV antibody product.
* Previous serious vaccine-associated AE or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including any wheezing event or reactive airway disease. Participants with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. Participants who had one episode of wheezing or received bronchodilator therapy for a single episode of illness in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months may also be enrolled.
* Member of a household that includes an immunocompromised individual or infants less than 6 months of age, other than a study participant
* Attends day care with infants less than 6 months of age, and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. Note: children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.

Inclusion Criteria for Seronegative Infants and Children:

* Healthy children at least 6 but less than 25 months of age whose parents/guardians can understand and sign the informed consent and who agree to vaccine administration following detailed explanation of the study
* Seronegative for RSV antibody, defined as a serum RSV neutralizing antibody titer less than 1:40 as determined not more than 42 days prior to inoculation
* Participant's history has been reviewed and participant has undergone a physical examination indicating that s/he is in good health. Permitted concomitant medications include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including topical steroids, topical antibiotics, and topical antifungal agents.
* Participant is expected to be available for the duration of the study

Exclusion Criteria for Seronegative Infants and Children:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy including systemic corticosteroids, or bone marrow/solid organ transplant recipients
* Major congenital malformations including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an RSV vaccine or previous receipt of or planned administration of any anti-RSV antibody product.
* Previous serious vaccine-associated AE or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including any wheezing event or reactive airway disease. Participants with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. Participants who had one episode of wheezing or received bronchodilator therapy for a single episode of illness in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months may also be enrolled.
* Member of a household that includes an immunocompromised individual or infants less than 6 months of age
* Attends daycare with infants less than 6 months of age, and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.

Inclusion Criteria for Infants (Group 4):

* Healthy infants 4 to 6 months of age whose parents/guardians can understand and sign the informed consent and who agree to vaccine administration following detailed explanation of the study.
* Subject's history has been reviewed and subject has undergone a physical examination indicating that s/he is in good health. Permitted concomitant medications include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including topical steroids, topical antibiotics, and topical antifungal agents.
* Subject is expected to be available for the duration of the study.

Exclusion Criteria for Infants (Group 4):

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy including systemic corticosteroids or bone marrow/solid organ transplant recipients.
* Major congenital malformations including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders.
* Previous immunization with an RSV vaccine or previous receipt of or planned administration of any anti-RSV antibody product.
* Previous serious vaccine-associated AE or anaphylactic reaction.
* Known hypersensitivity to any vaccine component.
* Lung or heart disease, including any wheezing event or reactive airway disease. Subjects with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled.
* Member of a household that includes an immunocompromised individual or infants less than 4 months of age.
* Attends daycare with infants less than 4 months of age, and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.

Temporary Exclusion Criteria for Seropositive Children, Seronegative Children, and Infants:

The following are temporary or self-limiting conditions, and once resolved, the subject may be enrolled, if otherwise eligible. If the period of temporary exclusion is greater than 42 days, seronegative children will need to be rescreened for levels of RSV neutralizing antibody.

* Fever (rectal temperature of greater than or equal to 100.4°F [38°C]), or upper respiratory illness (rhinorrhea, cough, or pharyngitis) or nasal congestion significant enough to interfere with successful vaccination, or otitis media
* Subject has received any killed vaccine or live attenuated rotavirus vaccine within 14 days prior to inoculation, any other live vaccine within 28 days prior to inoculation, or gamma globulin (or other antibody products) within the past 3 months prior to inoculation.
* Receipt of another investigational vaccine or investigational drug 28 days prior to receiving this investigational RSV vaccine
* Has received antibiotics or systemic or nasal steroid therapy for acute illness within the previous 3 days prior to vaccination (steroid skin creams or lotions and topical antibiotics or antifungal preparations are permitted)
* Has received salicylate (aspirin) or salicylate-containing products within 28 days prior to inoculation
* Children born at less than 37 weeks gestation and less than 1 year of age

Inclusion Criteria for Second Year of RSV Surveillance

* Those children who have completed the initial study and whose parents/guardians can understand and sign the informed consent.
* Subject is expected to be available during the second year of RSV surveillance.

Exclusion Criteria for Second Year of RSV Surveillance

* Currently enrolled in another RSV study.

Ages: 4 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of vaccine-related solicited adverse events (AEs) that occur during the intensive monitoring phase of the study | Measured at Days 0-10 for seropositive children and Days 0-28 for seronegative infants and children
Proportion of participants that develop 4-fold or greater rises in RSV neutralizing antibody titer following vaccination | Measured through follow-up period, up to 1 year after study entry
  Antibody responses to the RSV F glycoprotein will also be assessed by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research (CIR), Baltimore, Maryland
  - Center for Immunization Research South, Laurel, Maryland

REFERENCES:
- [Derived] Karron RA, Luongo C, Mateo JS, Wanionek K, Collins PL, Buchholz UJ. Safety and Immunogenicity of the Respiratory Syncytial Virus Vaccine RSV/DeltaNS2/Delta1313/I1314L in RSV-Seronegative Children. J Infect Dis. 2020 Jun 16;222(1):82-91. doi: 10.1093/infdis/jiz408. PMID 31605113